CLINICAL TRIAL: NCT02407535
Title: Assessing the Ultrasound Done on a the Uterus After Hysterectomy as a Diagnostic Tool for the Depth of Endometrial Carcinoma Invasion Into the Myometrium
Brief Title: Assessing Uterine Ultrasound Done as a Diagnostic Tool for the Depth of Carcinoma Invasion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Carmel Medical Center (Other)
Responsible Party: Principal Investigator, Ido Feferkorn, MD, Carmel Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CMC-14-0059-CTIL
Record Dates: First submitted 2015-03-12; First posted 2015-04-03 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Endometrial Endometroid Carcinoma

ARMS (1):
- Endometrial carcinoma patient (Experimental)
  Interventions: Device: Intraoperative ultrasound

INTERVENTIONS:
Device: Intraoperative ultrasound — Diagnostic intraoperative ultrasound in the uterus after hysterectomy for assessing depth of tumor invasion

SUMMARY:
In this study the investigators aim to assess the diagnostic performance of intraoperative, ultrasonographic assessment of the surgical extracted uterus for determining myometrial invasion's depth in comparison to preoperative ultrasound, intraoperative gross inspection and final pathological report (gold standard). The investigators hope that intraoperative gross inspection of the extracted uterus might offer an additional intraoperative tool for assessing the need for pelvic lymphadenectomy in early stage of endometrial cancer at least as good as pathological exam.

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age is 18 or above
2. Patient has been scheduled to undergo hysterectomy (laparoscopic or abdominal) for the staging and treatment of endometrial cancer (endometrioid subtype) and with the relevant suspected symptoms.
3. Patient able to understand,read and sign informed consent.
4. Patient is not participating in other medical trials at present or in the past 30 days

Exclusion Criteria:

1. Age under 18 years
2. Patients assessed preoperatively to be at stage 2 and higher endometrial carcinoma
3. Subjects which their biopsy in the pre operating process will include high risk cell types:

   * Grade 3 endometrioid adenocarcinoma,
   * clear cell carcinoma
   * papillary serous carcinoma
   * carcinosarcoma

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2015-03; Primary Completion 2018-06-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Tumor invasion | Average of 2 weeks (immediate assessment by ultrasound, average of 2 weeks for final pathological report)
  Tumor invasion (in millimeters and in percentage of myometrial size) as assessed by ultrasound in comparison to macroscopic assesment during surgery and to final pathological report)

CONTACTS AND LOCATIONS:
Overall Officials: Ido Feferkorn, MD, Principal Investigator — Carmel Medical Center
Locations (1):
- Carmel Medical Center, Haifa, Israel

IPD SHARING:
Plan to Share IPD: No